CLINICAL TRIAL: NCT01426945
Title: Evaluating Candidate Protein Expression in Human Rhabdomyosarcoma (RMS)
Brief Title: Protein Expression in Samples From Young Patients With Rhabdomyosarcoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ARST11B3; COG-ARST11B3 (Other: Children's Oncology Group); ARST11B3 (Other: Children's Oncology Group); NCI-2011-03534 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-08-31; First posted 2011-09-01 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Sarcoma
Keywords: alveolar childhood rhabdomyosarcoma; previously treated childhood rhabdomyosarcoma; previously untreated childhood rhabdomyosarcoma; recurrent childhood rhabdomyosarcoma; embryonal childhood rhabdomyosarcoma
MeSH Terms: conditions — Sarcoma | interventions — Immunohistochemistry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tumor tissue
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: protein expression analysis
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying tissue samples from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors find better ways to treat cancer.

PURPOSE: This research trial studies protein expression in samples from young patients with rhabdomyosarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To measure the protein expression of candidate proteins in human rhabdomyosarcoma (RMS) tumor samples.

OUTLINE: Archived tumor tissue samples are analyzed for protein expression (i.e., Notch1, Hey1, FGFR4, and Sp1) by IHC techniques and standard commercially available antibodies. Candidate proteins are then correlated with each patient age, gender, rhabdomyosarcoma (RMS) tumor stage, and RMS tumor subtype.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Tumor tissue samples from children with rhabdomyosarcoma (RMS) enrolled in the Children's Oncology Group clinical trials

  * Alveolar rhabdomyosarcoma (ARMS)
  * Embryonal rhabdomyosarcoma (ERMS)

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children with rhabdomyosarcoma (RMS) enrolled in the Children's Oncology Group clinical trials
Sampling Method: Non-Probability Sample
Enrollment: 77 (Estimated)
Dates: Start 2011-11; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
RMS protein expression profile

CONTACTS AND LOCATIONS:
Overall Officials: Corinne M. Linardic, MD, PhD, Principal Investigator — Duke Cancer Institute